CLINICAL TRIAL: NCT01148654
Title: Predicting Preterm Birth and Adverse Neonatal Outcomes With Novel Biomarkers: Identifying Those at Greatest Risk to Allow for Future Therapeutic Trials
Brief Title: The Biomarker Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Principal Investigator, Michal A. Elovitz, Associate Professor, Director, Maternal and Child Health Research Program, Department of Obstetrics and Gynecology, University of Pennsylvania
Other Study IDs: 807678
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Preterm Birth; Preterm Labor
Keywords: preterm birth; preterm labor; PTB; PTL
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal serum, plasma, saliva; Neonatal saliva

GROUPS / COHORTS (2):
- 1- Preterm Labor 22.0-33.6 weeks gestational age: Pregnant women between 22.0 and 33.6 weeks gestational age presenting to the Hospital of the University of Pennsylvania (HUP) complaining of Preterm labor (PTL), preterm premature rupture of membranes (PPROM), or cervical insufficiency (CI).
- 2- Preterm birth 34-36.6 weeks gestational age: Pregnant women delivering at the University of Pennsylvania between 34.0 and 36.6 weeks gestational age

SUMMARY:
Preterm birth (PTB) is a leading contributor to perinatal morbidity and mortality. While patients with preterm labor (PTL) are at an increased risk for PTB, not all PTL patients will deliver preterm. In patients with PTB, there is a high prevalence of 'intrauterine inflammation' as demonstrated by a large body of evidence. The presence of inflammation is noted by infiltration of inflammatory cells in the placenta and/or maternal fever in labor and/or elevation of cytokines in the amniotic fluid.

Despite this significant association of inflammation with PTB, identification of women destined to deliver preterm by inflammatory markers in maternal blood has not been successful. To date, it has been difficult to determine which patients with PTL will experience PTB. Identification of biomarkers, such as high sensitivity C-Reactive Protein (hsCRP) as well as others such as sICAM, Pentraxin, sE-Selectin, and CxCL-10 in maternal serum and in placental cord blood, may help to serve three very important clinical aims. 1) Identification of novel biomarkers in maternal serum could help to distinguish those women with PTL who are most likely to deliver PTB. 2) These biomarkers may have a high negative predictive value and thus identify those women who are not likely to deliver preterm, avoiding undue hospital admission and medical therapies. 3) Select biomarkers in the mother and/or in cord blood may serve to identify those preterm neonates at greatest risk for adverse outcome. Through improved identification of these infants, studies with targeted therapies to reduce adverse neonatal outcomes in preterm neonates become feasible.

This study involves a cohort assessment of women at risk for Preterm birth secondary to preterm labor, preterm premature rupture of membranes (PPROM), and cervical insufficiency (CI), between 22-0/7 and 33-6/7 weeks gestational age. We will obtain information regarding patients' pertinent past medical and obstetric history as well as small samples of maternal blood at up to four occasions, small samples of placental cord blood, a maternal saliva sample, and an infant buccal swab. We will follow each of these patient's pregnancy outcomes, and determine if there are any correlations between levels of certain biomarkers and latency to delivery as well as composite adverse neonatal outcomes. In women with PTB < 37 weeks, cord blood will be collected (as well as maternal saliva and an infant buccal swab) and biomarkers compared between those infants with and without specific adverse neonatal outcomes. Maternal saliva and buccal will be collected on all women and infants enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancies between 22-0/7 and 33-6/7 weeks gestational age who present to the Hospital of the University of Pennsylvania 'Perinatal Evaluation Center' (PEC) complaining of PTL, PPROM, or CI.
* Women who present to Labor and Delivery and will deliver (or have just delivered) a single infant preterm (22-0/7 to 36-6/7 weeks) at HUP.

Exclusion Criteria:

* Multiple-gestation, major fetal anomaly, fetal demise, severe preeclampsia prior to enrollment, patients on chronic steroid use or immunosuppressive drugs, patients with significant (active) immunological disease (AIDS, SLE), acute febrile illness (such as with active influenza or pyelonephritis), and pregestational diabetes.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with singleton pregnancies between 22-0/7 and 33-6/7 weeks gestational age who present to the Hospital of the University of Pennsylvania 'Perinatal Evaluation Center' (PEC) complaining of PTL, PPROM, or CI. Group 2: Women who present to Labor and Delivery and will deliver (or have just delivered) a single infant preterm (22-0/7 to 36-6/7 weeks) at HUP.
Sampling Method: Non-Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
preterm birth | enrollment through delivery

CONTACTS AND LOCATIONS:
Overall Officials: Michal A Elovitz, MD, Principal Investigator — University of Pennsylvania; Jamie A Bastek, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States